CLINICAL TRIAL: NCT04584034
Title: Bronchodilators for Wheeze in Young Children Presenting to Primary Care: a Randomised, Placebo-controlled, Multicentre, Parallel Group Trial
Acronym: KIWI
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Premature ending of the study due to impossibility of obtaining a suitable placebo-inhaler
Sponsor: UMC Utrecht (Other)
Collaborators: KU Leuven (Other); Maastricht University Medical Center (Other); Universiteit Antwerpen (Other); Université de Liège (Other)
Responsible Party: Principal Investigator, prof. dr. R.A.M.J. Damoiseaux, Full Professor, department of General Practice, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL72651
Record Dates: First submitted 2020-09-03; First posted 2020-10-12 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Wheezing
Keywords: Wheeze; Viral respiratory illnesses; Pre-school age children; Primary care; General practice; Salbutamol; Bronchodilators; Therapeutic trial
MeSH Terms: conditions — Respiratory Sounds | interventions — Albuterol; Bronchodilator Agents

STUDY DESIGN:
Intervention Model Description: Individually randomised, placebo-controlled, multicentre, parallel group trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Salbutamol (Active Comparator): Salbutamol inhalation 4x200ug daily for 7 days, delivered using a Babyhaler
  Interventions: Drug: Salbutamol
- Placebo (Placebo Comparator): Placebo 4 x 2 inhalations daily for 7 days, delivered using a Babyhaler
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Salbutamol — Salbutamol will be delivered using a Babyhaler spacer device. Ventolin will be used, brandname for Salbutamol sulfate. Ventolin contains the propellant HFA 134a.
  Other Names: Ventolin; β2-adrenoceptor agonist; Bronchodilator; Salbutamol sulfate
  Arms: Salbutamol
Drug: Placebo — The placebo will be delivered using a Babyhaler spacer device. The placebo will contain only the propellant HFA 134a.
  Other Names: Mock inhaler
  Arms: Placebo

SUMMARY:
Ten percent of infants are prescribed short-acting bronchodilators (i.e. salbutamol) for wheezing every year, yet evidence to support this treatment in children younger than two years old is scarce. The aim of this study is to evaluate the effectiveness and safety of salbutamol for treatment of wheezing in young children who present to their primary care physician.

In this study, the investigators will compare the effect of a 7-day treatment with salbutamol to the effect of 7-day treatment with a placebo. The main effect will be measured by evaluating a parent-reported symptom score. Additionally, the investigators will look at the presence of wheeze after 5 days, time to recovery, adverse events, healthcare utilisation, medication prescriptions, cost-effectiveness, and parent satisfaction with treatment.

DETAILED DESCRIPTION:
BACKGROUND: Worldwide, 30% of all infants and young children experience an episode of wheezing (Matricaldi et al. 2008; Mallol at al. 2010; Martinez et al. 1995). Currently, there is no evidence to underpin the management of these children. National Belgian and Dutch primary care professional guidelines propose 'a trial of treatment' with short acting bronchodilators (i.e. salbutamol) for wheezing children below the age of six years and to evaluate treatment effect after 1 to 2 weeks, but convincing evidence is lacking (Chavasse et al. 2002).

The effect of salbutamol has been studied well in children with proven asthma and is considered the first-line treatment in all patients in international asthma guidelines. However, trial findings of children with asthma are not applicable to primary care infants and young children with acute wheeze for several reasons; the anatomy and physiology in younger children differs significantly from those in older children and many infants and young children with an acute episode of wheezing do not experience further wheezing episodes later in life. As a result, it is at present unclear whether salbutamol inhalation therapy confers any benefit in young children who wheeze.

OBJECTIVE: To evaluate the (cost-)effectiveness of salbutamol inhalations (4x200μg for 7 days) versus placebo in children aged 6-24 months presenting to their primary care physician with wheezing.

DESIGN: A primary care based, randomised, placebo-controlled, multicentre, parallel group trial in 40 general practices and community paediatric practices in Belgium and the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to their primary care physician because of wheezing as confirmed by clinical examination (chest auscultation)
* A baseline score of 7 or higher on a parent-reported respiratory symptom score

Exclusion Criteria:

* Prematurity (<37 weeks)
* Major congenital malformations
* Pre-existing pulmonary disease as diagnosed by a paediatrician
* Continuous use of inhalation medication
* Physician visit because of wheezing in previous two weeks
* Use of inhalation medication in the previous two weeks
* Wheezing as a result of upper airway obstruction (i.e. laryngitis subglottica/pseudocroup)
* Severe illness requiring inhalation medication, prescription of antibiotics, or hospital referral during the consultation of inclusion

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Course of the parent reported respiratory symptom score | 5 days
  Scores on an arbitrary ordinal scale of 0 to 3 (0= no symptoms, 1= a bit (mild), 2= quite bad (moderate), 3= very bad (severe)) are recorded by parents for wheeze, cough and difficulty in breathing for both day and night, giving a maximum possible symptom score of 18 for each day.

SECONDARY OUTCOMES:
Time to recovery | 28 days
  Recovery defined as a respiratory symptom score of 5 or lower indicating only trivial symptoms
Adverse effects | 7 days
Health care resource use | 28 days
  Primary care physician re-consultations, medication prescriptions (e.g. antibiotics), specialist consultations and hospital admissions
Persistent wheezing on auscultation on day 5 | on day 5
  To maximise objectivity, lung sounds will be recorded (digital stethoscope) and evaluated by an expert panel at a later date
Day of parent reported recovery | 28 days
  The number of the day on which parents felt their child was recovered
Parent satisfaction with care | on day 28
  Single direct question "How satisfied are you with the treatment with study medication on a scale from 1 to 4 (very satisfied, satisfied, unsatisfied, very unsatisfied)?
Out-of-pocket expenses | 14 days
  Parent reported expenses for over-the-counter medication, additional travel, parking and child care, recorded in the study diary
Parent productivity losses | 14 days
  Assessed using the iMTA Productivity Cost questionnaire (iPCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Roger AMJ Damoiseaux, Professor, Principal Investigator — Julius Center, UMC Utrecht; Ann van den Bruel, Professor, Principal Investigator — KU Leuven

IPD SHARING:
Plan to Share IPD: Yes
We will make our data accessable for verification and future research (other researchers / spin-off projects), yet these will be shared under restrictions. Data cannot be reused without consulting the research team.
Time Frame: Data will only be accessable after publication of trial results. Data will be stored for at least 25 years.
Access Criteria: On request, after approval of principle investigator.

REFERENCES:
- [Background] Matricardi PM, Illi S, Gruber C, Keil T, Nickel R, Wahn U, Lau S. Wheezing in childhood: incidence, longitudinal patterns and factors predicting persistence. Eur Respir J. 2008 Sep;32(3):585-92. doi: 10.1183/09031936.00066307. Epub 2008 May 14. PMID 18480107
- [Background] Martinez FD, Wright AL, Taussig LM, Holberg CJ, Halonen M, Morgan WJ. Asthma and wheezing in the first six years of life. The Group Health Medical Associates. N Engl J Med. 1995 Jan 19;332(3):133-8. doi: 10.1056/NEJM199501193320301. PMID 7800004
- [Background] Mallol J, Garcia-Marcos L, Sole D, Brand P; EISL Study Group. International prevalence of recurrent wheezing during the first year of life: variability, treatment patterns and use of health resources. Thorax. 2010 Nov;65(11):1004-9. doi: 10.1136/thx.2009.115188. Epub 2010 Sep 20. PMID 20855440
- [Background] Chavasse R, Seddon P, Bara A, McKean M. Short acting beta agonists for recurrent wheeze in children under 2 years of age. Cochrane Database Syst Rev. 2002;2002(3):CD002873. doi: 10.1002/14651858.CD002873. PMID 12137663